CLINICAL TRIAL: NCT06525376
Title: Validity and Reliability of Smartphone Inclinometer Application for Measurement of Cervical Range of Motion: a Cross-sectional Study
Brief Title: Validity and Reliability of Smartphone Inclinometer Application for Measurement of Cervical Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Physical Therapy 2
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Joint Function Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: smartphone inclinometer application — an instrument for measuring angles of slope (or tilt), elevation, or depression of an object with respect to gravity.

SUMMARY:
Nowadays, smartphone technology provides opportunities for assessing and treating patients in clinical facilities and during the follow-up of the patient's progress. To date, many studies have assessed the validity and reliability of the smartphone application against universal goniometer for various joint motions, for instance, the spinal column, knee, and ankle. This study aims to determine the validity and reliability of smartphone inclinometer application for measurement of cervical region range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 33 years.
* Both genders.
* Subjects that are cooperative to follow my instructions

Exclusion Criteria:

* Subjects with severe spinal pathology.
* Pregnancy and lactation.
* Any musculoskeletal diseases that affect the cervical spine.
* Any neurological diseases that affect the cervical spine.
* History of trauma in the cervical spine.
* Signs of cervical radiculopathy.
* Signs of cervical myelopathy.
* Signs of serious pathology.
* subjects have a pacemaker or any other medical equipment that the magnet might have compromised.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Cervical range of motion device (CROM) | 6 weeks
  The cervical range of motion (ROM) serves as a functional measure of one's capacity for head and neck movement

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No